CLINICAL TRIAL: NCT00591058
Title: A Phase I Dose Escalation Study Evaluating the Safety and Biologically Active Dose of TM-601 Based on Perfusion MRI Imaging Criteria in Patients With Progressive and/or Recurrent Malignant Glioma
Brief Title: Safety and Dose-Finding Study of TM-601 in Adults With Recurrent Malignant Glioma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TransMolecular (Industry)
Responsible Party: TransMolecular, TransMolecular, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TM601-007
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; GBM; Astrocytoma; Oligodendroglioma
Keywords: recurrent glioma; Phase I; Multi-Center; Open label; Brain Cancer; Brain tumor; GBM; Glioma; Glioblastoma multiforme
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms | interventions — Chlorotoxin; Metabolism

ARMS (6):
- Cohort 1 (Experimental): 0.04 mg/kg TM-601 dose per administration
  Interventions: Drug: TM-601
- Cohort 2 (Experimental): 0.08 mg/kg TM-601 dose per administration
  Interventions: Drug: TM-601
- Cohort 3 (Experimental): 0.16 mg/kg TM-601 dose per administration
  Interventions: Drug: TM-601
- Cohort 4 (Experimental): 0.3 mg/kg TM-601 dose per administration
  Interventions: Drug: TM-601
- Cohort 5 (Experimental): 0.6 mg/kg TM-601 dose per administration
  Interventions: Drug: TM-601
- Cohort 6 (Experimental): 1.2 mg/kg TM-601 dose per administration
  Interventions: Drug: TM-601

INTERVENTIONS:
Drug: TM-601 — TM-601, administered intravenously (IV), once/week for 3 weeks
  Other Names: Chlorotoxin (Synthetic)

SUMMARY:
The purpose of this study is to evaluate the safety and biologically active dose of TM-601 in adult patients with recurrent malignant glioma.

DETAILED DESCRIPTION:
This Phase I study will evaluate the safety of TM-601 in patients with recurrent malignant glioma who have failed first-line, standard therapy.

Study patients will be assigned to receive treatment in 1 of 6 treatment cohorts. Patients will be assigned to each dose level in groups of 3-6 (depending upon treatment response seen within each cohort), with escalation to the next highest dose dependent upon demonstrated tolerance in the previous dosing group.

Patients will be administered an imaging dose of 131I-TM-601, intravenously, to demonstrate tumor-specific localization prior to study treatment with non-labeled TM-601. Eligible patients demonstrating tumor-specific imaging will be assigned to a treatment cohort and will received non-labeled TM-601 once a week for 3 weeks, followed by clinical follow-up visits and MR imaging.

Data from this study will help determine the IV dose of TM-601 required to produce MR perfusion changes (as well as other biomarker changes) in patients with recurrent malignant glioma. It is not known whether participation in this trial will provide patients with benefit in terms of improved tumor control, although pre-clinical evidence and evidence from other clinical trials with 131I TM-601 suggest that TM-601 is an active agent in malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

Patients Must:

1. Have histologically proven malignant glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or glioblastoma multiforme) which is progressive or recurrent after external beam radiation therapy (to at least 50 Gy) ± chemotherapy. Patients with previous low grade glioma who progressed after radiotherapy ± chemotherapy and are biopsied and found to have a high grade glioma are eligible.
2. Be ≥18 years of age.
3. Have a baseline Karnofsky Performance status of ≥60%
4. Have a Mini Mental State Exam score ≥ 19.
5. Have a life expectancy, based on the Investigator's judgment, of >3 months.
6. On screening ECG, have a QTc interval of <450 ms.
7. If taking steroids, be on a dose that is stable for at least 5 days prior to the imaging dose.
8. Have recovered from the toxicity of all previous therapy prior to enrollment. If the patient has undergone recent major surgery, an interval of at least 3 weeks must have elapsed between the surgery and the date of the imaging dose.
9. Have adequate organ and marrow function as defined below:

   hemoglobin >9.0g/dL absolute neutrophil count >1,500 mm3 platelet count >100,000 mm3 prothrombin time <1.5 ULN partial thromboplastin time (PTT) <1.5 ULN total bilirubin < 2.0 mg/dL AST(SGOT)/ALT(SGPT) <5 x institutional ULN creatinine (serum) ≤2.0 mg/dL*

   *If serum creatinine is >2.0 then creatinine clearance must be ≥60 ml/min
10. Have a negative serum and urine pregnancy test within 14 days of study drug administration, if female and of child bearing potential.
11. Agree to use an effective form of contraception to avoid pregnancy, if fertile (applicable to both male and female patients).
12. Agree to refrain from nursing, if female.
13. Have signed and dated written informed consent.
14. Be able to comply with treatment plan, study procedures and follow-up examinations.

Exclusion Criteria:

Patients may NOT:

1. Have a serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety. (Examples of medical illnesses are [but not limited to] the following: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.)
2. Have a prior malignancy with less than 5-year disease free interval, except for adequately treated basal cell or squamous cell carcinoma of the skin, or in situ cancer of the cervix.
3. Be pregnant or breast-feeding.
4. Have received radiation treatments ≤ 3 months from time of first study drug administration.
5. Have received any cytotoxic chemotherapy, whether conventional or investigational, ≤ 4 weeks prior to enrollment in this study (6 weeks for mitomycin-C or nitrosoureas).
6. Have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to 131I-TM-601 e.g. iodine or iodine-containing drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
To determine the safety profile/tolerability of TM-601 in this patient population, based on adverse event incidence, severity, duration, causality, seriousness and type as well as by physical examination, vital signs and clinical laboratory assessments. | Throughout the treatment phase of the study for each study patient, and for 28 days following the final study dose.

SECONDARY OUTCOMES:
A primary objective of this study is to evaluate the biologically active dose of TM-601 in this population of patients based on changes in perfusion MRI parameters. | At the completion of the dosing cycle for each patient, and at 28 days following the patient's final study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Burt Nabors, MD, Principal Investigator — University of Alabama at Birmingham; Glenn Lesser, MD, Principal Investigator — Wake Forest University; Steven Rosenfeld, MD, PhD, Principal Investigator — Columbia University; Sean Grimm, MD, Principal Investigator — Northwestern University; Maceij Mrugala, MD, Principal Investigator — University of Washington at Seattle; Jeremy Rudnick, MD, Principal Investigator — Cedars-Sinai Medical Center; Gerry Linette, MD, Principal Investigator — Washington University at St. Louis
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Mamelak AN, Jacoby DB. Targeted delivery of antitumoral therapy to glioma and other malignancies with synthetic chlorotoxin (TM-601). Expert Opin Drug Deliv. 2007 Mar;4(2):175-86. doi: 10.1517/17425247.4.2.175. PMID 17335414
- [Background] Mamelak AN, Rosenfeld S, Bucholz R, Raubitschek A, Nabors LB, Fiveash JB, Shen S, Khazaeli MB, Colcher D, Liu A, Osman M, Guthrie B, Schade-Bijur S, Hablitz DM, Alvarez VL, Gonda MA. Phase I single-dose study of intracavitary-administered iodine-131-TM-601 in adults with recurrent high-grade glioma. J Clin Oncol. 2006 Aug 1;24(22):3644-50. doi: 10.1200/JCO.2005.05.4569. PMID 16877732
- [Background] Hockaday DC, Shen S, Fiveash J, Raubitschek A, Colcher D, Liu A, Alvarez V, Mamelak AN. Imaging glioma extent with 131I-TM-601. J Nucl Med. 2005 Apr;46(4):580-6. PMID 15809479
- [Background] Lyons SA, O'Neal J, Sontheimer H. Chlorotoxin, a scorpion-derived peptide, specifically binds to gliomas and tumors of neuroectodermal origin. Glia. 2002 Aug;39(2):162-73. doi: 10.1002/glia.10083. PMID 12112367